CLINICAL TRIAL: NCT06354712
Title: Clinical Study Evaluating the Efficacy and Safety of N-acetylcysteine in Preventing Radiotherapy-Induced Oral Mucositis in Head and Neck Cancer Patients.
Brief Title: Efficacy of N-acetylcysteine in Preventing Radiotherapy-Induced Oral Mucositis in Head and Neck Cancer Patients.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Lecturer of Clinical Pharmacy and Pharmacy Practice, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-45
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Oral Mucositis (Ulcerative) Due to Radiation
Keywords: Oral Mucositis, Radiotherapy, N-acetylcysteine
MeSH Terms: conditions — Stomatitis; Ulcer | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Other): Standard Care
  Interventions: Drug: Institutional standard care
- Interventional arm (Active Comparator): Standard Care plus NAC
  Interventions: Drug: N-Acetyl-Cysteine with Institutional standard care

INTERVENTIONS:
Drug: N-Acetyl-Cysteine with Institutional standard care — A potent antioxidant and anti-inflammatory drug (A precursor of the endogenous antioxidant glutathione)
  Arms: Interventional arm
Drug: Institutional standard care — Benzydamine Mouthwash
  Arms: Control arm

SUMMARY:
A prospective, randomized, controlled, parallel clinical trial will be conducted at Clinical Oncology and Nuclear Medicine Center at Mansoura University Hospital to assess the efficacy of N-acetylcysteine in the prevention of radiotherapy induced oral mucositis in Head and Neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults >18 years diagnosed with squamous cell carcinoma of the head and neck scheduled to receive curative radiotherapy (Primary or postoperative) of at least 50 Gy with or without concurrent chemotherapy.
2. Individuals with healthy mucosa.
3. Adequate bone marrow function (Hemoglobin level ≥10 g/dL, platelet count ≥75 × 103/microliter, and absolute neutrophil count ≥1.5 × 103/microliter).
4. Patients with ECOG performance ≤2

Exclusion Criteria:

1. History of chemotherapy or radiotherapy.
2. Signs of systemic infections.
3. Pregnant and lactating women.
4. Individuals receiving systemic analgesics.
5. Liver disorders and renal failure with eGFR <30 ml/min/1.73m2 (by the MDRD equation).
6. Inability to follow instructions and complete the questionnaires.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of oral mucositis with grade ≥ 2 assessed weekly by World Health Organization scale for Oral Mucositis. | 8 weeks
  Difference between the two arms regarding incidence of grade ≥ 2 according to World Health Organization scale for Oral Mucositis.

SECONDARY OUTCOMES:
Time to develop oral mucositis with grade ≥ 2. | 8 weeks
  Difference between the two arms regarding time to develop oral mucositis with grade ≥ 2 according to WHO scale for oral mucositis.
  World Health Organization scale for oral mucositis
  * Grade 0: no oral mucositis
  * Grade 1: erythema and soreness
  * Grade 2: ulcers, able to eat solids
  * Grade 3: ulcers, requires liquid diet
  * Grade 4: ulcers, alimentation not possible (due to mucositis).
Duration of oral mucositis with grade ≥ 2. | 8 weeks
  Difference between the two arms regarding duration of oral mucositis with grade ≥ 2 according to WHO scale for oral mucositis.
Pain assessed by Visual Analog Scale (VAS). | 8 weeks
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression. The most simple VAS is a straight horizontal line of fixed length usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (worst) to the right (best).
  we will allocate this scale in comparing pain severity between the two arms.
Functional oral intake scale | 8 weeks
  TUBE DEPENDENT (levels 1-3)
  1. No oral intake
  2. Tube dependent with minimal/inconsistent oral intake 3 Tube supplements with consistent oral intake
  TOTAL ORAL INTAKE (levels 4-7) 4. Total oral intake of a single consistency 5. Total oral intake of multiple consistencies requiring special preparation 6. Total oral intake with no special preparation, but must avoid specific foods or liquid items 7. Total oral intake with no restrictions
Patient's quality of life assessed by Functional Assessment of Cancer Therapy in Head and Neck Cancer (FACT-H&N) version 4 | 8 weeks
  A questionnaire filled by head and neck cancer patient to assess the quality of life.
  H&N1 I am able to eat the foods that I like H&N2 My mouth is dry H&N3 I have trouble breathing H&N4 My voice has its usual quality and strength H&N5 I am able to eat as much food as I want H&N6 I am unhappy with how my face and neck look H&N7 I can swallow naturally and easily H&N8 I smoke cigarettes or other tobacco products H&N9 I drink alcohol (e.g. beer, wine, etc.) H&N10 I am able to communicate with others H&N11 I can eat solid foods H&N12 I have pain in my mouth, throat or neck
  Scoring:Not at all (0) A little bit (1) Somewhat (2) Quite a bit (3) Very much(4)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed el-Husseiny shams, Professor, Principal Investigator — Department of Clinical pharmacy and Pharmacy practice, Faculty of Pharmacy, Mansoura University; Noha Mansour, phD, Study Director — Department of Clinical pharmacy and Pharmacy practice, Faculty of Pharmacy, Mansoura University; Rasha Mohamed Abd-Ellatif, Professor, Study Director — Center of Clinical Oncology and nuclear medicine, Faculty of Medicine, Mansoura University; Fatma Gharib Khirallah, Associate Professor, Study Director — Center of Clinical Oncology and nuclear medicine, Faculty of Medicine, Tanta University; Mohamed Awad Ebrahim, Professor, Study Director — Center of Medical Oncology and Adult BMT, Faculty of Medicine, Mansoura University.
Locations (1):
- Clinical Oncology and Nuclear Medicine of Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided